CLINICAL TRIAL: NCT00149617
Title: Career Training in Marijuana Dependence
Brief Title: Effectiveness of Buspirone and Motivational Enhancement Therapy for the Treatment of Marijuana Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Aimee L. McRae, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-15440-1; K23DA015440 (NIH); K23-15440-1; DPMC
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2007-12

CONDITIONS: Marijuana Abuse; Mood Disorders
Keywords: Marijuana; Mood Disorder
MeSH Terms: conditions — Marijuana Abuse; Mood Disorders | interventions — Buspirone

INTERVENTIONS:
Drug: Buspirone

SUMMARY:
This study will assess the effectiveness of a combination of buspirone and motivational interviewing therapy in the treatment of marijuana dependence.

DETAILED DESCRIPTION:
Marijuana dependence is one of the most common substance-related disorders in the United States. Despite its prevalence, there is a lack of clinical research addressing treatments for marijuana dependence. Research has shown that marijuana abuse is associated with affective disorders. This may be caused by repeated use for relief from anxiety. The use of an anxiolytic agent, a drug that relieves anxiety, may help treat marijuana dependence. Motivational enhancement therapy has been shown to reduce marijuana use. Therefore, it is likely that buspirone, which is an anxiolytic agent, combined with motivational enhancement therapy will prove beneficial in treating marijuana dependence. This study will assess the effectiveness of a combination of buspirone and motivational interviewing in the treatment of marijuana dependence.

This double-blind study will last a total of 16 weeks. Participants will be randomly assigned to receive either buspirone or placebo for a period of 12 weeks. There will be one follow-up appointment 4 weeks post-intervention. Baseline assessments will include a physical exam and urine and blood tests. Study visits will occur weekly throughout treatment in order to monitor compliance, assess adverse affects, and obtain substance use data. Mood assessment scales, marijuana craving questionnaires, and a withdrawal symptom checklist will be used to gather the data. Urine drug screens will be collected weekly to test for marijuana use. In addition to this, the presence of opioids, cocaine, amphetamines, and benzodiazepines will be tested at baseline, Weeks 6 and 12, and at follow-up. A 10-day supply of medication will be dispensed to participants each week. Meetings for motivational enhancement therapy will last 30 to 90 minutes each and will occur at baseline, Week 2, and Week 4. Participants' perceived quality of life will be measured at baseline and Weeks 6 and 12 to determine the effect of buspirone.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for marijuana dependence
* Lives within 60 miles of the study site
* Willing to provide collateral individuals for contact purposes
* Willing to use an effective form of contraception throughout the study

Exclusion Criteria:

* Meets DSM-IV criteria for dependence upon a substance other than marijuana, nicotine, or caffeine
* Meets DSM-IV criteria for a history of schizophrenia or another non-affective psychotic disorder or bipolar disorder
* Meets DSM-IV criteria for current major depressive disorder or eating disorder
* Significant cognitive impairment
* Currently taking benzodiazepines, antidepressant, or antipsychotic medications
* Major medical illnesses (e.g., HIV, kidney failure, unstable angina, chronic obstructive pulmonary disease, infectious hepatitis)
* Not in stable housing
* Pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2004-04; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Drug use; measured at Weeks 12 and 16

SECONDARY OUTCOMES:
Anxiety; measured at Week 12
Craving; measured at Week 12
Withdrawal symptoms; measured at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Mcrae, Pharm.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States